CLINICAL TRIAL: NCT02933307
Title: Continuous Monitoring of Vital Signs in Hospitalized Patients
Brief Title: Continuous Monitoring on the General Ward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HEEL-2015-03
Record Dates: First submitted 2016-07-25; First posted 2016-10-14 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2016-07

CONDITIONS: Carcinoma, Pancreatic Ductal; Colorectal Neoplasms; Arthritis; Hypertension; Sepsis
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal; Colorectal Neoplasms; Arthritis; Hypertension; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention): Patients with regular measurements by nurses only (Modified Early Warning Score (MEWS))
- HealthPatch (Intervention) (Experimental): Patients with HealthPatch and regular MEWS measurements
  Interventions: Device: HealthPatch
- ViSi Mobile (Intervention) (Experimental): Patients with ViSi Mobile and regular MEWS measurements
  Interventions: Device: ViSi Mobile

INTERVENTIONS:
Device: HealthPatch — The HealthPatch (Vital Connect) is a wireless patch and continuously measures single-lead ECG, heart rate, respiratory rate, stress, skin temperature, body posture and steps
  Arms: HealthPatch (Intervention)
Device: ViSi Mobile — ViSi Mobile (Sotera Wireless) is wireless device that is able to continuously measure all important vital parameters: ECG, heart rate, oxygen saturation, blood pressure, respiratory rate and skin temperature.
  Arms: ViSi Mobile (Intervention)

SUMMARY:
Rationale: Monitoring patients' vital signs is done to detect clinical deterioration. For this, the MEWS, a scoring list comprising seven vital signs measured by nursing staff, is used. Although the MEWS provides relevant data on patients' health status, the interval measurements may not capture early deterioration of vital signs, especially during the night. As a result, unsafe situations may occur such as periods of low oxygen saturation and cardiac arrhythmias, which are known to complicate postoperative course. Besides, this way of measuring vital signs may be stressful for patients and disturbs patients' sleep. New technology such as ViSi Mobile and HealthPatch allows for remote continuous monitoring of vital signs using wearable devices transmitting relevant data to nurses and clinicians. With this, the investigators think that clinical deterioration may be detected in an early phase and reduce nurse work load and patient distress.

Objective: to investigate the feasibility of wearable devices on the general ward.

Study design: feasibility study.

Study population: adult patients hospitalized on the internal medicine ward and adult postoperative patients on the surgical ward.

Intervention: patients in the intervention groups will be randomized in one of the two groups. Patients in the group 1 will wear ViSi Mobile; patients in group 2 will wear the HealthPatch. Wearable devices will be worn for at least three days. Regular MEWS measurements take place at usual time points.

Main study parameters/endpoints: Evaluation with patient and care givers (primary outcome measure), MEWS calculations, time between alarm (continuous data) and next regular MEWS measurement (nurse), intervention by nurse after alarm, admission to ICU, complications, side effects of devices, STAI scores, and PCS scores will be documented.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients will wear one device for at least three days. Devices can be uncomfortable by being heavy or the patches can start itching. More measurements by nurses can take place when indicated, for example after alarms. The participating patients will fill out the STAI on daily basis and the PCS on the last day of hospitalization. Both questionnaires will take a few minutes to complete. Patients could benefit from early detection of clinical deterioration and early corrective interventions or ICU admissions.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years or older on the day the informed consent will be signed.
* Patient is hospitalized on the surgical or internal medicine ward.
* MEWS measurements are required at least three times a day.
* Patient is able to speak, read and understand the local language of the investigational site, is familiar with the procedures of the study, and agrees to participate in the study program by giving oral and written informed consent prior to screening evaluations.

Exclusion Criteria:

* Frequency of MEWS measurements is less than three times a day.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Expectations & experiences of patients | 2-3 days after informed consent
  Interviews of 15-20 minutes with patients after 2-3 days wearing a device or control group
Expectations & experiences of care givers | 1 year
  Interviews with nurses of 15-20 minutes at the end of the study. Estimated amount of 6 nurses

SECONDARY OUTCOMES:
MEWS scores based on continuous data and data measured by nurses | 3 times a day, up to three days.
Amount of alarms by HealthPatch or ViSi Mobile | during 2-3 days when the patient wears a device
Time between alarm (continuous data) and next regular MEWS measurement (nurse) | during 2-3 days when the patient wears a device
Amount of extra MEWS measurements by nurses due to alarms | during 2-3 days when the patient wears a device
Admission to ICU (yes/no) | during 2-3 days when the patient participates in this study
Duration of ICU hospitalization in days | during 2-3 days when the patient participates in this study
Complications caused by disease or surgical procedure | during 2-3 days when the patient participates in this study
Adverse events caused by devices | during 2-3 days when the patient wears a device
  E.g. Itch or redness
Technical failures of devices (artifacts: a period longer than 1 minute the device does not measure vital parameters) | during 2-3 days when the patient wears a device
Outcomes of the State Trait Anxiety Inventory (STAI) | Once a day during the 2-3 days the patient participantes in this study
Outcomes of the Pain Catastrophizing Scale (PCS) | On day 2 or 3 when patients participates in the study
System usability Scale | 1 year

OTHER OUTCOMES:
Gender | On day 1 when patients participates in the study
  Extraction from EHR
Age | On day 1 when patients participates in the study
  Extraction from EHR
Diagnosis | On day 1 when patients participates in the study
  Extraction from EHR
Performed surgical procedure | On day 1 when patients participates in the study
  Extraction from EHR

CONTACTS AND LOCATIONS:
Overall Officials: Harry van Goor, MD, PhD, FRCS, Principal Investigator — Radboud University Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weenk M, Bredie SJ, Koeneman M, Hesselink G, van Goor H, van de Belt TH. Continuous Monitoring of Vital Signs in the General Ward Using Wearable Devices: Randomized Controlled Trial. J Med Internet Res. 2020 Jun 10;22(6):e15471. doi: 10.2196/15471. PMID 32519972